CLINICAL TRIAL: NCT07371546
Title: Continuous Glucose Monitoring (CGM) in Prediabetes: A Mixed-Methods Study Exploring Behavioural Impact, Patient Experiences and Provider Perspectives
Brief Title: Continuous Glucose Monitoring (CGM) in Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0022-APP1
Record Dates: First submitted 2025-06-23; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pre-diabetes
Keywords: Primary care; Continuous glucose monitoring; Behavioural change; Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Participants in the intervention arm will wear the Abbott Freestyle Libre system for 2 weeks, in addition to usual care.
  Interventions: Device: Continuous Glucose Monitoring
- Control (No Intervention)

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Participants will also receive the Abbott Freestyle Libre system, which is a sensor-based flash glucose monitoring system that has been approved by the U.S. Food and Drug Administration for personal use by patients since September 2017 (Office of the Commissioner, 2020). Participants will also receive device-specific education and be taught how they can use CGM data to identify foods or physical activities more likely to affect their glucose levels.
  Arms: Intervention

SUMMARY:
Part 1 and 2 of study (For Patient Participants) The purpose of this study is to examine if the wearing of a medical device called a continuous glucose monitor (CGM) can guide adults with prediabetes modify their behaviors and manage their health, compared to traditional health coaching. Prediabetes means the study participants have a higher-than-normal blood sugar level which is not high enough to be considered type 2 diabetes yet but will put them at risk of developing it. CGM measures glucose levels without the participants having to prick fingers and involves wearing a small sensor on the back of the arm day and night which allows viewing of glucose levels on the mobile phone with a painless 1 second scan.

This is the first time the investigators are trying to do research using CGM for adults with prediabetes. the study team want to learn how practical it is to do such a study. The study will explore if wearing of a CGM sensor makes a difference in terms of health outcomes compared to regular health coaching. It also aims to understand the users' experience with the CGM system.

This study targets to recruit 76 participants from Pasir Ris Polyclinic.

Part 1 of the study uses a research method called a randomized controlled trial. Participants who consent to join will be allocated to one of two groups based on chance. Half of the participants will receive the CGM sensor in addition to health coaching. This is called the intervention group. The other half of the participants will receive health coaching alone. This is called the control group. Participants in both groups will continue regular follow-up with their own primary care physicians.

There will be 3 study touchpoints, which will mainly be at Pasir Ris Polyclinic.

1. Baseline visit:

   * Receive health coaching that will take 20-30 minutes.
   * Complete questionnaires about socio-demographic details, diet and physical activity which will take 20-30 minutes.
   * Measure weight, body mass index (BMI), and waist circumference.
   * Past medical history and medications will be retrieved from the electronic medical records.
   * If the participants are in the intervention group, the study team will assist them to apply the Abbott Freestyle Libre continuous glucose monitoring (CGM) sensor and link it to their smartphone. The study team will also set up the LibreLink app and Libreview account.
2. 1-month touchpoint

   * Complete follow up questionnaires to assess any changes in the diet and physical activity.
   * This touchpoint may be conducted either face-to-face or via a phone call.
3. 6-month touchpoint

   * Complete final questionnaires about the lifestyle.
   * Measure weight, BMI and waist circumference again
   * Uninstall the LibreLink app and Libreview account.

Part 2 of the study is an in-depth interview to understand the experiences of the participants using the Abbott Freestyle Libre CGM System. This part of the study will be conducted either during the 3rd study touchpoint or on another day (within 9 months from start of intervention). The interview will last 60 minutes and will be audio-recorded. Questions asked will be regarding the general experience using the CGM, any difficulties with following the study instructions and suggestions to improve the study.

Part 3 of study for Healthcare Providers Participants (HCP):

The purpose of this study is to assess the effects of CGM on adults with prediabetes and to explore the facilitators and barriers of using CGM in prediabetes management from both patients and healthcare providers. The study aims to understand the perspectives of primary care providers on the potential benefits, challenges, and feasibility of integrating CGM into prediabetes management. The findings will help pave the way for broader integration of CGM technology into public health programs targeting specific populations at high risk of diabetes to improve health outcomes.

If the participants agree to participate, they will be invited to fill in a data collection form on the demographics, qualifications and clinical experience. This will take 20-30 minutes. The participants will be interviewed either individually or in a group with other of their colleagues from the same polyclinic. During the interview, the researcher will ask questions pertaining to their experiences with prediabetes management, knowledge of CGM and their views of the potential challenges and opportunities in the utilization of CGM by prediabetic adults. The interviews will be audio recorded. participation in the study will last approximately 60 minutes.

DETAILED DESCRIPTION:
BACKGROUND The World Health Organization (WHO) has identified diabetes as a priority non-communicable disease and launched initiatives to promote its prevention and management. Type-2 diabetes mellitus (T2DM) account for 90% of all global diabetes cases. Many countries have implemented national screening programs for early interventions and mitigate the associated complications. Such screening programs result in identifying people with pre-diabetes, a dysglycemic state in which the individuals are at increased risks of developing T2DM. Pre-diabetes include those with impaired glucose tolerance (IGT) or impaired fasting glucose (IFG) or both IGT and IFG. At least 35% of individuals with pre-diabetes will progress to T2DM within eight years without lifestyle changes. Individuals with prediabetes also have an increased risk of developing microvascular and macrovascular complications, even before progressing to frank T2DM.

The global prevalence of IGT and IFG in 2021 was 9.1% (464 million) and 5.8% ((298 million) respectively and is expected to rise to 638 million in 2045. The prevalence of prediabetes is highest in developed countries. Singapore is no exception; 14% of its adult population being identified with prediabetes.

Pre-diabetes opens a window for early intervention to de-escalate the progression to T2DM. Lifestyle interventions such as diet or exercise for adults with prediabetes can effectively mitigate their dysglycemia. A meta-analysis on pooled results from eleven randomized controlled trials reported that individuals with prediabetes who underwent lifestyle interventions had 36% lower risk of progressing to T2DM, resulting in significant gains in their quality adjusted life-years. In the Diabetes Prevention Program, the incidence of T2DM was reduced by 34% with lifestyle modifications and 18% with metformin at the 10-year follow-up. However, the potential success of effective lifestyle modifications is diluted by difficulties in adherence to healthy behaviors.

Failure to control pre-diabetes is multi-factorial. At the individual level, people with pre-diabetes lack understanding of their glycemic state and are unaware of the dietary and lifestyle measures to prevent its deterioration. They have limited access to interventions in structured programs, and do not receive adequate follow-up care or support after their diagnosis, leading to inaction. At the system level, traditional diets high in refined carbohydrates and unhealthy cooking can be difficult to modify. Social gatherings and workplace environments may also discourage healthy behaviors. The rising prevalence of obesity, sedentary lifestyle and unhealthy diets have contributed to the increasing failure to control pre-diabetes. Harnessing medical technology to enhance self-efficacy in pre-diabetes management is an option to overcome these multi-faceted barriers.

Existing tools such as continuous glucose monitoring (CGM) has been shown to improve diabetes care by providing direct and timely feedback to patients with T1DM or T2DM on their meal-related glycemic fluctuations. It is preferred over traditional capillary blood glucose monitoring due to convenience, comfort and ease of use. CGM has been deployed in prediabetes in small-scale studies in the United States of America and Canada, which reported that its short-term use in adults increased their adherence to lifestyle interventions, such as reducing food portion sizes, choosing healthier food alternatives, and increasing physical activity levels. Subsequently, the Asia-Pacific Diabetes Care Advisory Board in 2021 has recommended individuals with prediabetes to leverage on CGM to gather constant feedback on their glycemic status and to motivate their behavioral change.

Aligned with the recommendations, the Health Promotion Board in Singapore has recently launched a community-based program which aims to use CGM as one of the prediabetes interventions to improve health outcomes. However, the effectiveness and efficacy of using CGM to modify lifestyle and dietary behavior among adults with pre-diabetes, compared to routine diabetic counselling or health coaching have yet to be elucidated.

AIMS The overarching aim of the study is to assess the impact of CGM in modifying the lifestyles of adults with prediabetes. Specifically, the study primarily aims to determine the effectiveness of CGM in raising their diabetes literacy, adopting low carbohydrate and fat diet, increasing their frequency and intensities of physical activities, reducing their weight, body mass index and waist circumference over a period of 24-28 weeks.

The study also aims to

1. Explore and understand the facilitators and barriers of using CGM in prediabetes management from the key stakeholders, including both the individuals and their clinicians.
2. Determine if trial design was appropriate and was feasible with regards to i) subject recruitment and retention ii) adherence to protocol, iii) adverse events iii) patient acceptability of the intervention before planning a full scale randomized controlled trial.

   METHODS This study is a mixed-method study conducted at Pasir Ris Polyclinic. It is expected to take 18 months to complete. The first part of the study is a pilot two-armed, randomized controlled trial. The second part of the study involves in-depth interviews with the intervention arm participants. The third part of the study involves interviews with the healthcare providers. Due to the nature of the intervention, only the outcome assessors are blinded.

   Sample Size Part 1 (Pilot randomized controlled trial) The sample size calculation is based on sample size recommendation to use at least 30 subjects or greater to estimate a parameter in a pilot study. Assuming that the main trial is to be designed with 90% power and two-sided 5% significance, a pilot trial sample size per treatment arm of 25 and more will detect a small, standardized effect size that is around 0.2. The sample size will take into account possible 20% drop out, hence the final sample size is increased to 38 per arm (n=76).

   Part 2 and 3 (Qualitative interviews) In this qualitative part of the study, sample size is determined by data saturation, which is reached when additional data no longer reveal new themes or insights. Different guidelines exist for determining sample size for qualitative research. Bertaux (1981) proposed 15 as the smallest accepted sample. Creswell and Poth (2016) recommended 20-30 interviews to be sufficient while Morse (2000) suggested 30 as an estimated number to reach theoretical saturation. Therefore, the sample size for part 2 and 3 of the study will be a maximum of 30 patients and 30 healthcare providers respectively.

   Recruitment and Sampling Part 1 and 2 Recruitment of participants will be done by convenient sampling. Primary Care Physicians and Healthcare workers in Pasir Ris Polyclinic will be engaged to help identify suitable patients. Eligible patients will be verbally asked by their attending physicians to participate in the study. If the participants agree to participate, the attending doctor will complete the consultation. After doctor consultation, participants will be directed to the study team to check for eligibility, briefed on the purpose of the study and obtain written informed consent. The study procedures will be administered during the same visit. Subjects who require time to consider will be provided with the participant information sheet to read through at leisure. They will be invited to return another day if agreeable to participate and written consent will be obtained by the study team.

   The participants will be randomly assigned to either the intervention or control group in a 1:1 ratio according to a pre-defined computer-generated sequence using the permuted blocks randomization technique. This predefined sequence of numbers will be concealed in sequentially numbered, sealed, opaque envelopes. Envelopes are opened after eligibility has been confirmed and written informed consent obtained.

   Participants in the intervention arm will be asked at point of recruitment if they consent to take part in the interview. They will be briefed on the purpose of the study, their roles, their rights and that the interview will be digitally audio recorded. If agreeable, they will proceed with the interviews after de-identification. The expected participation time is 60 minutes.

   Part 3 The healthcare providers (HCP) caring for the participants that will be recruited. include primary care physicians, nurses and clinicians from other domains who have provided direct care to adults with prediabetes.. They will be invited to participate at the end of clinic meetings. Potential participants not present at the clinic meetings will be contacted by the study team in person. Written consent will be obtained from the healthcare providers who agree to participate in the qualitative interview. The expected participation time is 60 minutes.

   Participants will be reimbursed with a voucher (SGD 20) at each of the three touchpoints for the first part of the study. Participants who complete part 2 of the study will be given an additional voucher of SGD 20. Healthcare providers who agree to partake in part 3 of the study will be reimbursed with SGD 20.

   Part 1 (Pilot randomized controlled trial) All participants will have 3 study touchpoints at baseline (week 0), week 2-6 and week 24-28. At week 0, a healthcare professional will individually go through a prediabetes health education slide deck with participants from the control and intervention arms. The slide deck was developed by Singhealth Polyclinics in 2022, and includes topics on the pathophysiology and complications of pre-diabetes, diabetes risk assessment, and non-pharmacological management of the condition. After the health education, participants will be asked to list the food types and physical activities they feel are likely to affect glycemic control, and encouraged to make necessary lifestyle modifications.

   At the baseline week 0 visit, participants randomized to the intervention group will receive the Abbot Freestyle Libre system. The study team will assist the participants in applying the sensors and setting up their LibreLink app and LibreView accounts. Each participant will register for the accounts using a unique participant code as their user ID, an email address generated by the research team, and their LibreView accounts will be linked to the Principal Investigator's account. The unblinded sensor will be activated and linked to the participant's smartphone, and the participant will receive device-specific education. Participants in this group will be instructed to scan their glucose levels every 8 hourly at a minimum but can choose to scan more frequently. They will also be taught how to make diet and activity modifications to limit glucose excursions above 7.8 mmol/l, and how they could use CGM data to identify foods or physical activities more likely to affect their glucose levels, especially the ones they have listed earlier. The study team will help the participants to uninstall their LibreLink apps and Libreview accounts at the 3rd study touchpoint.

   Questionnaires are administered at each of the three touchpoints. These touchpoints will be conducted be face-to-face at Pasir Ris Polyclinic. The questionnaire includes the thirty-seven-item diet screener (DS) and International Physical Activity Questionnaire-Short Form for diet and physical activity measures respectively. Waist circumference, weight, and Body Mass Index (BMI) are measured at baseline and at week 24-28.

   Participants from the intervention and control arms will receive standard care from their physicians, and any medication titration is left to the discretion of the physicians during routine follow-up.

   Part 2 (In-depth interviews with the intervention arm participants) On the 3rd visit touchpoint, participants in the intervention group who have earlier consented for this part of the study will undergo in-depth interviews conducted in a quiet room at Pasir Ris Polyclinic. If the participants are unable to complete the interviews at the third study touchpoint, they may reschedule for another day, provided that all interviews are conducted within 36 weeks from the start of the intervention. The first interview will be overseen by a study team member with qualitative research experience. The principal investigator/co-investigators will conduct the interviews. The interviews are audio-recorded, and live transcription will will be transcribed verbatim using the research department's transcribing software, transcription platforms (such as transcribe.gov.sg or Note Buddy) or engagement of professional transcribers.

   Part 3 (Interviews/ focus group discussions with the healthcare providers) Part 3 of the study will run concurrently with part 1. Healthcare providers who cared for adults with prediabetes and consented to be interviewed will undergo either in-depth interviews or partake in a focus group discussion. This will be conducted in-person, in a quiet room at Pasir Ris Polyclinic. The first interview will be overseen by a study team member with qualitative research experience. The principal investigator/co-investigators will conduct the interviews. The interviews are audio-recorded, and live transcription will be performed with an artificial intelligence transcription tool.

   Research Instruments Baseline Measures

   The following baseline data will be collected at the 1st study touchpoint for all participants:
   1. Sociodemographic data, including year of birth, gender, ethnic group, marital status, occupational status, education level and current housing type
   2. Risk factors for diabetes - family history of diabetes, history of gestational diabetes, smoking
   3. Co-morbidities, duration of prediabetes, metformin use (electronic medical records)
   4. Measurements of body weight, body mass index (BMI), waist circumference
   5. 37-item Diet Screener
   6. International Physical Activity Questionnaire Short Form

   Sociodemographic data for HCPs The data collected from HCPs include age, gender, ethnic group, qualifications, years of practice and job title.

   Qualitative interview topic guides Topic guides will be used during the in-depth interviews/ focus group discussions

   For the intervention arm participants, it will cover four main segments: (1) general experience in using CGM; (2) challenges, constraints, potential advantages of utilising CGM; (3) the facilitators and barriers to lifestyle behavioral change with the interventions; (4) recommendations for improvement of the study procedures.

   For the HCPs, the following questions will be explored: (1) experience with managing adults with prediabetes; (2) knowledge and experience with CGM; (3) views on using CGM in adults with prediabetes; (4) facilitators and barriers to offering CGM as part of prediabetes management to their patients.

   Data Collection For quantitative data, we will use REDCAP, a database management system to capture research data electronically. It is a secure web application for building and managing databases.

   Participants' LibreView accounts will be linked to the Principal Investigator's account, allowing for secure and centralized data access to the glucose data for research purposes by the study team members.

   For qualitative data, audio recording of the interviews will be by digital voice recorder. We will be using the research department's transcribing software, transcription platforms (such as transcribe.gov.sg or Note Buddy) or engagement of professional transcribers. All identifiable information in the transcripts will be removed before analysis.

   Medical Device:

   Abbott Freestyle Libre Glucose Monitoring System and LibreLink App.

   FreeStyle LibreLink app ('App') when used with a FreeStyle Libre Flash Glucose Monitoring System Sensor ('Sensor') measures interstitial fluid glucose levels in people (age 4 and older). The App and Sensor are designed to replace blood glucose testing in the self-management of diabetes, including dosing of insulin but has been used in research and in diabetes prevention program in people who are normoglycemia or have prediabetes. It has been registered locally with Health Sciences Authority.

   The study team members will be trained in the proper administration of the device by other study team members familiar with its application in regular clinical practice. They will help the participants administer the sensors during the first study visit and dispose of the sensor applicators at the clinic. Participants will be taught how to remove it themselves after 14 days and dispose of it via standard waste collection. The device is only administered once in the study and participants are not required to re-administer it at home.

   Participants will register for LibreLink app and LibreView accounts using a unique participant code as their user ID and an email address generated by the research team. Participants' LibreView accounts will be linked to the Principal Investigator's account, allowing for secure and centralized data access to the glucose data for research purposes by the study team members.

   Data Analysis Quantitative Descriptive statistics will be generated for the baseline characteristics of the study participants, and frequencies and percentages will be presented for categorical variables while mean and standard deviation will be presented for continuous variables. Normality of the continuous variables will be assessed using the Shapiro-Wilk test, and non-normal variables will be presented in median and interquartile ranges.

   Comparison of body weight, BMI, waist circumference, DS scores and MET at baseline between CGM and non-CGM group will be assessed using independent t-test if the variables are normally distributed, and Mann-Whitney U test if they are skewed.

   General estimating equation will be performed to examine the longitudinal time points for each outcome, using Intervention as the main covariate, and baseline characteristics as other covariates. All analyses will be analyzed using IBM SPSS version 29.0 and Stata MP version 18.5. A p-value of 0.05 is considered statistically significant.

   Qualitative Recording will be transcribed by a digital scribe or professional transcribers. Transcription will be audited and coded by at least 2 independent study team members. Thematic analysis will be performed after familiarization with the data. After completion of open coding from the first 3 in-depth interviews using grounded theory approach, consensus on the coding framework will be reached between study team members. This framework will then be applied to the subsequent interviews and codes expanded or modified after each deliberation. In the event of discrepancies in the coding framework among the study team members, this will be resolved through consensus.

   The data will be coded using the NVivo-12 software.

ELIGIBILITY:
Patient Participants

Inclusion Criteria:

1. Singaporean Citizen or Permanent Resident
2. Age 21 - 69 years old
3. Clinical diagnosis of prediabetes defined as a fasting glucose of 6.1-6.9 mmol/L and/or 2-hour glucose level of 7.8-11.0 mmol/L after an oral glucose tolerance test (Appropriate Care Guide, 2021)

   a. Can be conservatively managed, or medically managed with metformin
4. Owns a mobile phone that can download the Singapore FreeStyle LibreLink App
5. Expressed willingness to use participate in the study, use the devices according to the study protocol during the study period, and to sign informed consent.

Exclusion Criteria:

1. Pregnant or planned pregnancy within the next six months
2. Physical limitation that prevents the patient from engaging in physical exercise
3. Cognitively impaired based on diagnosis of dementia or mild cognitive impairment (MCI) in the electronic health records (EHR)
4. Not adequately proficient in English
5. Currently enrolled in another study or program that involves weight loss or dietary modifications, or novel therapeutic drug or device
6. Planned surgery in the next six months
7. Not able to use smartphone or the Singapore FreeStyle LibreLink App despite coaching
8. Any end-stage disease with life prognosis of < 2 years
9. Patients who are not willing or are not able to commit to the entire study program

Healthcare Providers (HCP) Participants HCPs from Pasir Ris Polyclinic who self-reported to have treated adults with prediabetes will be enrolled for the interviews.

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | 0 weeks, 2-6 weeks, 24-28 weeks
  37-item Diet Screener (DS) The DS was designed and validated in a multi-ethnic population locally aged 18-79 years to assess intakes of selected food groups that could represent overall dietary patterns. The screener covers intakes of whole grains, soya protein, fruit, vegetables, oily fish and dairy fat and demonstrates reasonably good validity and reproducibility relative to the more accepted but longer 163-item Food Frequency Questionnaire. It is therefore easier to administer during the study with minimal participant burden.
Physical activity using International Physical Activity Questionnaire Short Form | 0 weeks, 2-6 weeks, 24-28 weeks
  a validated 7-item instrument that measures an individual's physical activity in the last 7 days; measures metabolic equivalent of task (MET)-minutes per week. Participants are asked to report the days and time they spent in the last 7 days in 4 categories: vigorous activity (heavy lifting, aerobics, fast bicycling), moderate activity (light lifting, moderate bicycling), walking, and sitting (watching TV, reading). The total physical activity was calculated as the sum of the vigorous, moderate, and walking categories in metabolic equivalent minutes per week (MET-min per week scores). Questions on sitting are related to sedentariness and are scored separately. MET minutes represent the amount of energy expended carrying out physical activity. One MET is what the participants expend when they rest. To get a continuous variable score it is considered walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS. Higher score, better outcome.
Body weight | 0 week, 24-28 weeks
  Weight in kilograms
Height | 0 week, 24-28 weeks
  Height in meters
Body Mass Index | 0 week, 24-28 weeks
  Weight and Height will be combined to report Body Mass Index in kg/m^2
Waist circumference | 0 week, 24-28 weeks
  Waist circumference in centimeters: Waist circumference is measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest with a measuring tape. The mean value of two waist circumference measurements is used. Both measurements are repeated if there is a difference of more than 1 cm.

SECONDARY OUTCOMES:
Participant recruitment numbers | 6 months recruitment period
  Number of participants recruited for the control and intervention arm. The study targets to recruit 76 participants over a 6-month recruitment period.
Drop-out rate | 18 months study duration
  Number of participants that dropped out of the study. Drop-out rate is calculated based on the proportion of enrolled participants who do not complete the intervention/1-month follow-up/6-month follow-up. The study targets for a drop-out rate of < 20%.
Adherence rate to the sensor | 2-6 weeks
  Intervention group participants usage of CGM over the two-week period. Statistics on sensor adherence will be obtained from the Abbott Freestyle Libre system and is determined as >70% CGM use in the 2 weeks it is worn (≥10 readings over 2 weeks).
Exploring views on the facilitators and barriers of behavioral change with CGM | 24-28 weeks, to allow up to 36 weeks
  In-depth interviews with the intervention group participants
Views and experiences of using CGM with the Abbott Freestyle Libre system | 24-28 weeks, to allow up to 36 weeks
  In-depth interviews with the intervention group participants
Views and experiences on the study protocol | 24-28 weeks, to allow up to 36 weeks
  In-depth interviews with the intervention group participants
Experiences with managing adults with prediabetes | Baseline, up to 60 minutes
  Interviews with HCP participants till point of data saturation
Knowledge and experience with CGM | Baseline, up to 60 minutes
  Interviews with HCP participants till point of data saturation
Views on using CGM in adults with prediabetes | Baseline, up to 60 minutes
  Interviews with HCP participants till point of data saturation
Facilitators and barriers to offering CGM as part of prediabetes management to their patients | Baseline, up to 60 minutes
  Interviews with HCP participants till point of data saturation

OTHER OUTCOMES:
CGM data | 2-6 weeks
  Clinical CGM metrics extracted will consist of percentage of time CGM is active, number of glucose readings in 2 weeks, average glucose, time in range (TIR) of 3.9 to 10 mmol/l, time in tight range (TITR) of 3.9-7.8 mmol/l, time above range > 7.8 mmol/l (%TAR 7.8 mmol/l), time above range >10 mmol/l (%TAR 10 mmol/l), glycemic variability (GV, as standard deviation [SD] and the coefficient of variation [CV]) (Battelino et al., 2023).
No of participants with reportable adverse outcomes | 2-6 weeks
  All device or study-related adverse events, and sensor insertion or sensor wear-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jun Lim, BScHons, MD, Principal Investigator — SingHealth Polyclinics
Locations (1):
- Pasir Ris Polyclinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The patient consent forms have not included permission for broad data sharing or secondary analyses. There are also concerns about maintaining participant confidentiality and data privacy, as the study involves sensitive health information and is conducted in a clinical setting and data sharing could increase the risk of re-identification despite de-identification measures.

REFERENCES:
- [Background] Yadav R, Jain N, Raizada N, Jhamb R, Rohatgi J, Madhu SV. Prevalence of diabetes related vascular complications in subjects with normal glucose tolerance, prediabetes, newly detected diabetes and known diabetes. Diabetes Metab Syndr. 2021 Sep-Oct;15(5):102226. doi: 10.1016/j.dsx.2021.102226. Epub 2021 Jul 20. PMID 34303917
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Unger J, Kushner P, Anderson JE. Practical guidance for using the FreeStyle Libre flash continuous glucose monitoring in primary care. Postgrad Med. 2020 May;132(4):305-313. doi: 10.1080/00325481.2020.1744393. Epub 2020 Mar 30. PMID 32223687
- [Background] Schmidt K, Faerch K, Zoffmann V, Amadid H, Varming AR. The process of health behaviour change following participation in a randomised controlled trial targeting prediabetes: A qualitative study. Diabet Med. 2022 Apr;39(4):e14748. doi: 10.1111/dme.14748. Epub 2021 Dec 7. PMID 34806793
- [Background] Rooney MR, Fang M, Ogurtsova K, Ozkan B, Echouffo-Tcheugui JB, Boyko EJ, Magliano DJ, Selvin E. Global Prevalence of Prediabetes. Diabetes Care. 2023 Jul 1;46(7):1388-1394. doi: 10.2337/dc22-2376. PMID 37196350
- [Background] Richardson KM, Schembre SM, da Silva V, Blew RM, Behrens N, Roe DJ, Marvasti FF, Hingle M. Adding a Brief Continuous Glucose Monitoring Intervention to the National Diabetes Prevention Program: A Multimethod Feasibility Study. J Diabetes Res. 2024 May 16;2024:7687694. doi: 10.1155/2024/7687694. eCollection 2024. PMID 38919262
- [Background] Palladino R, Tabak AG, Khunti K, Valabhji J, Majeed A, Millett C, Vamos EP. Association between pre-diabetes and microvascular and macrovascular disease in newly diagnosed type 2 diabetes. BMJ Open Diabetes Res Care. 2020 Apr;8(1):e001061. doi: 10.1136/bmjdrc-2019-001061. PMID 32332069
- [Background] Morse, J. M. (2000). Determining Sample Size. Qualitative Health Research, 10(1), 3-5.
- [Background] Lim RBT, Wee WK, For WC, Ananthanarayanan JA, Soh YH, Goh LML, Tham DKT, Wong ML. Correlates, Facilitators and Barriers of Healthy Eating Among Primary Care Patients with Prediabetes in Singapore-A Mixed Methods Approach. Nutrients. 2019 May 6;11(5):1014. doi: 10.3390/nu11051014. PMID 31064063
- [Background] Lee JY, Nguyen JT, Arroyo J, Tran T, Hanami D, Mayorga J. Feasibility and Acceptability of Using Flash Glucose Monitoring System Sensors to Empower Lifestyle Changes in People With Prediabetes. Diabetes Care. 2023 Jan 1;46(1):e10-e11. doi: 10.2337/dc22-0612. No abstract available. PMID 36398782
- [Background] Kerrison G, Gillis RB, Jiwani SI, Alzahrani Q, Kok S, Harding SE, Shaw I, Adams GG. The Effectiveness of Lifestyle Adaptation for the Prevention of Prediabetes in Adults: A Systematic Review. J Diabetes Res. 2017;2017:8493145. doi: 10.1155/2017/8493145. Epub 2017 Apr 16. PMID 28567425
- [Background] IPAQ Group. (2005, November). Guidelines for data processing and analysis of the international physical activity questionnaire (IPAQ_-short and long forms. (2005).
- [Background] Health Promotion Board. (2024, November 14). HEALTH PROMOTION BOARD COLLABORATES WITH TECHNOLOGY AND HEALTHCARE PARTNERS TO INCUBATE SOLUTIONS THAT WILL HELP SINGAPOREANS PREVENT AND MANAGE CHRONIC CONDITIONS. Health Promotion Board
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] How Many Interviews Are Enough?: An Experiment with Data Saturation and Variability Greg Guest, Arwen Bunce, and Laura JohnsonView all authors and affiliations Volume 18, Issue 1
- [Background] Glechner A, Keuchel L, Affengruber L, Titscher V, Sommer I, Matyas N, Wagner G, Kien C, Klerings I, Gartlehner G. Effects of lifestyle changes on adults with prediabetes: A systematic review and meta-analysis. Prim Care Diabetes. 2018 Oct;12(5):393-408. doi: 10.1016/j.pcd.2018.07.003. Epub 2018 Aug 1. PMID 30076075
- [Background] Qualitative inquiry and research design: Choosing among five approaches. JW Creswell, CN Poth - 2016
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Carlson AL, Mullen DM, Bergenstal RM. Clinical Use of Continuous Glucose Monitoring in Adults with Type 2 Diabetes. Diabetes Technol Ther. 2017 May;19(S2):S4-S11. doi: 10.1089/dia.2017.0024. PMID 28541137
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Bertaux, D. (1981). From the life-history approach to the transformation of sociological practice. In Biography and society: The life history approach in the social sciences (pp. 29-45). London : Sage.
- [Background] Beaglehole R, Bonita R, Horton R, Adams C, Alleyne G, Asaria P, Baugh V, Bekedam H, Billo N, Casswell S, Cecchini M, Colagiuri R, Colagiuri S, Collins T, Ebrahim S, Engelgau M, Galea G, Gaziano T, Geneau R, Haines A, Hospedales J, Jha P, Keeling A, Leeder S, Lincoln P, McKee M, Mackay J, Magnusson R, Moodie R, Mwatsama M, Nishtar S, Norrving B, Patterson D, Piot P, Ralston J, Rani M, Reddy KS, Sassi F, Sheron N, Stuckler D, Suh I, Torode J, Varghese C, Watt J; Lancet NCD Action Group; NCD Alliance. Priority actions for the non-communicable disease crisis. Lancet. 2011 Apr 23;377(9775):1438-47. doi: 10.1016/S0140-6736(11)60393-0. Epub 2011 Apr 5. PMID 21474174
- [Background] Battelino T, Alexander CM, Amiel SA, Arreaza-Rubin G, Beck RW, Bergenstal RM, Buckingham BA, Carroll J, Ceriello A, Chow E, Choudhary P, Close K, Danne T, Dutta S, Gabbay R, Garg S, Heverly J, Hirsch IB, Kader T, Kenney J, Kovatchev B, Laffel L, Maahs D, Mathieu C, Mauricio D, Nimri R, Nishimura R, Scharf M, Del Prato S, Renard E, Rosenstock J, Saboo B, Ueki K, Umpierrez GE, Weinzimer SA, Phillip M. Continuous glucose monitoring and metrics for clinical trials: an international consensus statement. Lancet Diabetes Endocrinol. 2023 Jan;11(1):42-57. doi: 10.1016/S2213-8587(22)00319-9. Epub 2022 Dec 6. PMID 36493795
- [Background] Bailey KJ, Little JP, Jung ME. Self-Monitoring Using Continuous Glucose Monitors with Real-Time Feedback Improves Exercise Adherence in Individuals with Impaired Blood Glucose: A Pilot Study. Diabetes Technol Ther. 2016 Mar;18(3):185-93. doi: 10.1089/dia.2015.0285. Epub 2016 Feb 17. PMID 26885934
- [Background] Appropriate Care Guide. (2021). Agency for Care Effectiveness (ACE). Managing pre-diabetes - a growing health concern. Ministry of Health, Singapore. go.gov.sg/acg-managing-pre-diabetes-a-growing-health-concern